CLINICAL TRIAL: NCT03404570
Title: A Double-Blind, Randomized, Placebo-Controlled Exploratory Study to Assess the Efficacy and Safety of TC-5214 in the Treatment of Subjects With Moderate to Severe Palmar Hyperhidrosis
Brief Title: Exploratory Study to Assess the Efficacy and Safety of TC-5214 in the Treatment of Subjects With Palmar Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atacama Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-9951-201
Record Dates: First submitted 2017-12-22; First posted 2018-01-19 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Palmar Hyperhidrosis
Keywords: Sweaty Hands

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized (1:1:1) to one of three Treatment Arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study drug will be provided as oral tablets with active and placebo indistinguishable in product and packing characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose (4 mg) (Experimental): Oral tablet containing 2 mg of active drug, dexmecamylamine HCl. Subjects will be instructed to take two tablets by mouth once daily (in the morning).
  Interventions: Drug: Dexmecamylamine HCl
- Low Dose (2 mg) (Experimental): Oral tablet containing 1 mg of active drug, dexmecamylamine HCl. Subjects will be instructed to take two tablets by mouth once daily (in the morning).
  Interventions: Drug: Dexmecamylamine HCl
- Placebo (Placebo Comparator): Oral tablet containing no active drug. Subjects will be instructed to take two tablets by mouth once daily (in the morning).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmecamylamine HCl — Investigational drug
  Other Names: TC-5214
  Arms: High Dose (4 mg); Low Dose (2 mg)
Other: Placebo — Oral tablet containing no active drug.
  Arms: Placebo

SUMMARY:
This is a pilot exploratory study to evaluate the safety and efficacy of TC-5214 in subjects with palmar hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of primary hyperhidrosis of the palms
* Subject is currently drug-naïve for hyperhidrosis medications
* Females must be post-menopausal, surgically sterile, or use an effective method of birth control.

Exclusion Criteria:

* Subject is pregnant, lactating, is planning to become pregnant during the study, or is less than one year postpartum.
* Subject is a smoker within one year prior to Visit 1/Screening.
* Subject has known history of secondary hyperhidrosis.
* Subject has existence of neurological, psychiatric, endocrine, or other disease that can cause secondary hyperhidrosis or affect sweating.
* Subject has known history of Sjögren's syndrome or Sicca syndrome.
* Subject has used any of the following hyperhidrosis medications or therapies within the specified timeframe:

  1. Iontophoresis to the palms within four weeks prior to baseline visit;
  2. Botulinum toxin to the palms within one year prior to baseline visit;
  3. Prior surgical procedures to the palms (e.g., sympathectomy, debulking of sweat glands);
  4. Prior medical device treatment to the palms (approved or investigational);
  5. Any treatments for hyperhidrosis within four weeks prior to baseline visit.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has previously participated in a clinical study of dexmecamylamine or TC-5214.
* Subject has used an investigational drug or investigational device treatment within 30 days prior to baseline.
* Subject has a history of sensitivity to any of the ingredients in the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
HDSS Success | Day 14 (End of Treatment)
  Proportion of subjects with at least a 1, 2, or 3 point reduction in Hyperhidrosis Disease Severity Scale (HDSS) score from Baseline

SECONDARY OUTCOMES:
Reduction in Sweat Production | Day 14 (End of Treatment)
  Proportion of subjects with a ≥50% reduction in gravimetrically measured sweat production
Absolute change of Sweat Production | Day 14 (End of Treatment)
  Absolute change from Baseline in gravimetrically measured sweat production.

OTHER OUTCOMES:
Number of Subjects with Adverse Events (AEs) | From Baseline (Day 1) to End of Study (Day 22)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Site 02, San Diego, California
  - Site 03, St Louis, Missouri
  - Site 01, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No